CLINICAL TRIAL: NCT01986790
Title: Effective Communication to Improve Decision Making About Health Care Plans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HS020309
Record Dates: First submitted 2013-11-04; First posted 2013-11-18 (Estimated); Results first posted 2016-06-09 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-05

CONDITIONS: Health Literacy; Health Insurance; Health Services Accessibility
Keywords: Health insurance; Health services accessibility; Decision making; Health literacy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Plain Language (Experimental): This intervention group will receive a plain-language table describing the features and costs of health insurance plans, with definitions of health insurance terms incorporated into the table.
  Interventions: Behavioral: Plain Language
- Plain Language + Visuals (Experimental): This intervention group will receive the plain-language table plus visuals that focus on specific features of the plans. Participants will be able to view the information about each health insurance feature one feature at a time, in the order they prefer.
  Interventions: Behavioral: Plain Language + Visuals
- Plain Language + Narratives (Experimental): This intervention group will receive the plain language table plus narratives about how others might use and rate the insurance plans.
  Interventions: Behavioral: Plain Language + Narratives

INTERVENTIONS:
Behavioral: Plain Language
  Arms: Plain Language
Behavioral: Plain Language + Visuals
  Arms: Plain Language + Visuals
Behavioral: Plain Language + Narratives
  Arms: Plain Language + Narratives

SUMMARY:
The overall goal of the study is to better understand how communication strategies can help people make decisions about health insurance plans.

This study aims to:

* (Aim 1) Examine currently uninsured individuals' understanding of terminology and details of health insurance plans;
* (Aim 2) Apply three recommended strategies for communicating information about health insurance plans;
* (Aim 3) Test the effects of these strategies in a randomized experiment.

DETAILED DESCRIPTION:
First, this study will examine people's understanding of health insurance plan terminology and details through qualitative interviews with 50 uninsured individuals. These responses will then lead to the development of three communication strategies to improve understanding of health insurance plans: 1) plain language, 2) plain language plus visual displays and 3) plain language plus narratives.

The strategies will the be pilot tested with 30 individuals to assess readability, clarity of language, and layout. The revised communication strategies will be tested with 280 individuals in a randomized experiment. Individuals will be randomly assigned to either a plain language condition alone, a plain language + visual displays condition, and a plain language + narrative condition.

ELIGIBILITY:
Inclusion Criteria:

* Must be without health insurance currently
* Must have been without health insurance at some point in the past 12 months
* Must speak English

Exclusion Criteria:

* Currently has health insurance and has not had any lapses in coverage in the past 12 months
* Does not speak English

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 343 (Actual)
Dates: Start 2012-04; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Politi, PhD, Principal Investigator — The Washington University in St. Louis School of Medicine
Locations (1):
- The Washington University in St. Louis School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Gold M, Wooldridge J. Surveying consumer satisfaction to assess managed-care quality: current practices. Health Care Financ Rev. 1995 Summer;16(4):155-73. PMID 10151887
- [Background] Harris-Kojetin LD, McCormack LA, Jael EF, Sangl JA, Garfinkel SA. Creating more effective health plan quality reports for consumers: lessons from a synthesis of qualitative testing. Health Serv Res. 2001 Jul;36(3):447-76. PMID 11482584
- [Background] Hibbard JH, Jewett JJ, Engelmann S, Tusler M. Can Medicare beneficiaries make informed choices? Health Aff (Millwood). 1998 Nov-Dec;17(6):181-93. doi: 10.1377/hlthaff.17.6.181. PMID 9916368
- [Background] Peters E, Dieckmann N, Dixon A, Hibbard JH, Mertz CK. Less is more in presenting quality information to consumers. Med Care Res Rev. 2007 Apr;64(2):169-90. doi: 10.1177/10775587070640020301. PMID 17406019
- [Background] Hibbard JH, Slovic P, Jewett JJ. Informing consumer decisions in health care: implications from decision-making research. Milbank Q. 1997;75(3):395-414. doi: 10.1111/1468-0009.00061. PMID 9290635
- [Background] Knutson DJ, Kind EA, Fowles JB, Adlis S. Impact of report cards on employees: a natural experiment. Health Care Financ Rev. 1998 Fall;20(1):5-27. PMID 10387425
- [Background] Scanlon DP, Chernew M, Lave JR. Consumer health plan choice: current knowledge and future directions. Annu Rev Public Health. 1997;18:507-28. doi: 10.1146/annurev.publhealth.18.1.507. PMID 9143729
- [Background] Kreuter MW, Green MC, Cappella JN, Slater MD, Wise ME, Storey D, Clark EM, O'Keefe DJ, Erwin DO, Holmes K, Hinyard LJ, Houston T, Woolley S. Narrative communication in cancer prevention and control: a framework to guide research and application. Ann Behav Med. 2007 Jun;33(3):221-35. doi: 10.1007/BF02879904. PMID 17600449
- [Background] McCormack LA, Uhrig JD. How does beneficiary knowledge of the Medicare program vary by type of insurance? Med Care. 2003 Aug;41(8):972-8. doi: 10.1097/00005650-200308000-00010. PMID 12886176
- [Background] Hoadley J. Medicare Part D: simplifying the program and improving the value of information for beneficiaries. Issue Brief (Commonw Fund). 2008 May;39:1-15. PMID 18536148
- [Background] Lubalin JS, Harris-Kojetin LD. What do consumers want and need to know in making health care choices? Med Care Res Rev. 1999;56 Suppl 1:67-102; discussion 103-12. doi: 10.1177/1077558799056001S04. PMID 10354679
- [Background] Kolstad JT, Chernew ME. Quality and consumer decision making in the market for health insurance and health care services. Med Care Res Rev. 2009 Feb;66(1 Suppl):28S-52S. doi: 10.1177/1077558708325887. Epub 2008 Nov 24. PMID 19029288
- [Background] Hibbard JH, Jewett JJ. Will quality report cards help consumers? Health Aff (Millwood). 1997 May-Jun;16(3):218-28. doi: 10.1377/hlthaff.16.3.218. PMID 9141339
- [Background] Uhrig JD, Harris-Kojetin L, Bann C, Kuo TM. Do content and format affect older consumers' use of comparative information in a Medicare health plan choice? Results from a controlled experiment. Med Care Res Rev. 2006 Dec;63(6):701-18. doi: 10.1177/1077558706293636. PMID 17099122
- [Background] Kreuter MW, Wray RJ. Tailored and targeted health communication: strategies for enhancing information relevance. Am J Health Behav. 2003 Nov-Dec;27 Suppl 3:S227-32. doi: 10.5993/ajhb.27.1.s3.6. PMID 14672383
- [Background] Hinyard LJ, Kreuter MW. Using narrative communication as a tool for health behavior change: a conceptual, theoretical, and empirical overview. Health Educ Behav. 2007 Oct;34(5):777-92. doi: 10.1177/1090198106291963. Epub 2006 Dec 15. PMID 17200094
- [Background] Hibbard JH, Peters E. Supporting informed consumer health care decisions: data presentation approaches that facilitate the use of information in choice. Annu Rev Public Health. 2003;24:413-33. doi: 10.1146/annurev.publhealth.24.100901.141005. Epub 2001 Nov 6. PMID 12428034
- [Background] Politi MC, Kaphingst KA, Kreuter M, Shacham E, Lovell MC, McBride T. Knowledge of health insurance terminology and details among the uninsured. Med Care Res Rev. 2014 Feb;71(1):85-98. doi: 10.1177/1077558713505327. Epub 2013 Oct 24. PMID 24163306
- [Derived] Politi MC, Kaphingst KA, Liu JE, Perkins H, Furtado K, Kreuter MW, Shacham E, McBride T. A Randomized Trial Examining Three Strategies for Supporting Health Insurance Decisions among the Uninsured. Med Decis Making. 2016 Oct;36(7):911-22. doi: 10.1177/0272989X15578635. Epub 2015 Apr 3. PMID 25840904

RESULTS

PARTICIPANT FLOW:
Groups:
- Plain Language: This intervention group will receive a plain-language table describing the features and costs of health insurance plans, with definitions of health insurance terms incorporated into the table.
  Plain Language
- Plain Language + Visuals: This intervention group will receive the plain-language table plus visuals that focus on specific features of the plans. Participants will be able to view the information about each health insurance feature one feature at a time, in the order they prefer.
  Plain Language + Visuals
- Plain Language + Narratives: This intervention group will receive the plain language table plus narratives about how others might use and rate the insurance plans.
  Plain Language + Narratives
Period: Overall Study
Arm/Group | Plain Language | Plain Language + Visuals | Plain Language + Narratives
Started | 91 | 154 | 98
Completed | 91 | 154 | 98
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Plain Language | Plain Language + Visuals | Plain Language + Narratives | Total
Number analyzed (Participants) | 91 | 154 | 98 | 343
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.9 (12.0) | 38.7 (11.7) | 37.8 (12.1) | 38.5 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 79 | 63 | 203
  Male | 30 | 75 | 35 | 140
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 1 | 7
  Not Hispanic or Latino | 80 | 136 | 88 | 304
  Unknown or Not Reported | 9 | 14 | 9 | 32
Race/Ethnicity, Customized [Number; unit: Participants]
  African American | 48 | 87 | 59 | 194
  White | 31 | 42 | 24 | 97
  Other | 5 | 11 | 6 | 22
  Not Reported | 7 | 14 | 9 | 30
Region of Enrollment [Number; unit: Participants]
  United States | 91 | 154 | 98 | 343
Rapid Estimate of Adult Literacy in Medicine-SF (REALM-SF) [Number; unit: Participants] — Health literacy was assessed by the REALM-SF. 9th grade reading level or above=adequate, 7th or 8th grade reading level=marginal, 6th grade reading level or below=inadequate.
  Participants
    Inadequate | 6 | 11 | 8 | 25
    Marginal | 31 | 56 | 42 | 129
    Adequate | 52 | 85 | 44 | 181
    Not Reported | 2 | 2 | 4 | 8
Subjective Numeracy Scale (SNS) [Mean (Standard Deviation); unit: Units on a scale] — Subjective numeracy was measured using the validated Subjective Numeracy ability subscale. All questions were scored as marked (range 1-6), using the average rating across all 4 questions. A higher value is considered to be a better outcome.
  Units on a scale | 4.1 (1.1) | 4.2 (1.0) | 3.7 (1.2) | 4.0 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Knowledge
Description: Knowledge measures the degree at which participants understand the details about health insurance plans. Knowledge was scored on a scale from 0 to 7 based on number of correct answers to the 7 items. A higher value is considered to be a better outcome. Bivariate outcome data can be found below.
Time Frame: 1 day (Immediately following showing the participant the assigned intervention (plain language table, plain language table + visuals, or plain language table + narratives)
Population: Analysis is represented as mean (standard deviation) of calculated knowledge.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Plain Language | Plain Language + Visuals | Plain Language + Narratives
Number analyzed (Participants) | 91 | 154 | 98
Units on a scale | 6.0 (1.2) | 5.7 (1.3) | 5.5 (1.5)

2. Primary Outcome: Uncertainty
Description: A survey will be administered in order to measure participants' confidence in the features of health insurance plans that matter most to them and the insurance plan they chose of the ones presented. Confidence in choice is scored on a scale from 0 to 100, with higher scores indicating more decisional conflict/more uncertainty/less confidence in choice. Bivariate outcome data can be found below.
Time Frame: as for outcome 1
Population: Analysis is represented as mean (standard deviation) of calculated uncertainty.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Plain Language | Plain Language + Visuals | Plain Language + Narratives
Number analyzed (Participants) | 91 | 154 | 98
Units on a scale | 9.6 (21.6) | 10.6 (23.3) | 7.2 (18.8)

3. Primary Outcome: Satisfaction
Description: A survey will be administered in order to measure the extent to which participants are satisfied with the information presented to them. Satisfaction was scored on a scale from 1 to 4, with higher scores indicating higher levels of satisfaction. Bivariate outcome data can be found below.
Time Frame: as for outcome 1
Population: Analysis is represented as mean (standard deviation) of calculated satisfaction.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Plain Language | Plain Language + Visuals | Plain Language + Narratives
Number analyzed (Participants) | 91 | 154 | 98
Units on a scale | 2.7 (0.5) | 2.6 (0.5) | 2.7 (0.4)

ADVERSE EVENTS:
Description: "Serious" and "Other" adverse events were not collected/assessed.
Arm/Group | Plain Language | Plain Language + Visuals | Plain Language + Narratives
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No